CLINICAL TRIAL: NCT04383587
Title: Seroprevalence of SARS CoV 2 Antibodies in Previously Undiagnosed Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark A. Parkulo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-004054
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: SARS-CoV 2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serologic Arm (Other): Enrolled participants will have COVID19 IgG antibody testing performed.
  Interventions: Other: Serologic testing

INTERVENTIONS:
Other: Serologic testing — COVID19 IgG antibody testing to be performed

SUMMARY:
The purpose of this study is to identify healthcare workers with SARS CoV 2 antibodies who have not been previously diagnosed and are presumed COVID-19 negative, then determine the level of immunity in this population which could inform further decisions about widespread antibody testing in a healthcare worker population.

DETAILED DESCRIPTION:
Enrolled participants will complete a survey gauging their level of confidence they will be antibody positive. Participants will then complete serologic testing for SARS CoV 2 IgG antibodies. The study will characterize the prevalence of antibody positivity in this population and assess whether there is a correlation between a pre-test confidence level using a Likert scale and actual antibody positivity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Mayo Clinic employee in procedural and surgical area.
* Suspected COVID-19 exposure.
* Completed PCR test twice with negative results.

Exclusion Criteria:

- Refusal to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Parkulo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 394 invited to participate. 300 elected to participate. 292 completed study.
Groups:
- Serologic Arm: Enrolled participants will have COVID19 IgG antibody testing performed.
  Serologic testing: COVID19 IgG antibody testing performed
Period: Overall Study
Arm/Group | Serologic Arm
Started | 300
Completed | 292
Not Completed | 8

BASELINE CHARACTERISTICS:
Groups:
- Serology Group: Group of participants completing COVID Serologic antibody testing
Arm/Group | Serology Group
Number analyzed (Participants) | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 284
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 43 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174
  Male | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 292

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With COVID-19 Antibodies
Description: Presence of IgG antibodies detected
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Serologic Arm
Number analyzed (Participants) | 292
Participants
  Positive Antibodies | 8
  Negative Antibodies | 284
Statistical Analysis 1: Comparison: Serologic Arm; Participants were grouped by age (18-35 vs. 36-50 vs. 51-65 vs. >65), Sex at birth (Female vs. Male). and Occupational Role (Technician vs Anesthesiologist vs Advanced Practice Provider vs. Attendant Aide vs. CRNA vs. OR nurse vs Perfusionist vs Surgeon); Test type: Superiority; p > 0.18, Fisher Exact

2. Secondary Outcome: Ability to Predict Immune Status/Antibody Positivity
Description: Survey of participants to gauge their confidence they will be antibody positive
Time Frame: Single point in time prior to COVID-19 Antibody testing
Population: Of 292 participants completing the study, 27 responded in a survey (prior to antibody testing) that they had a high confidence (8 or greater on a Likert Scale from 0-10) that they had been previously infected with SARS CoV-2 and would test COVID-19 antibody positive. Antibody results from those 27 participants are listed below.
Measure: Count of Participants; unit: Participants
Groups:
- High Confidence of Previous Infection: Participants who indicated in a survey prior to antibody testing that they had a high confidence of previous infection or immunity that would be demonstrated by antibody positivity
Arm/Group | High Confidence of Previous Infection
Number analyzed (Participants) | 27
Participants
  Antibody negative | 26
  Antibody positive | 1

ADVERSE EVENTS:
Time Frame: Participants were instructed to contact investigators if they developed any adverse events within 1 week of blood draw.
Description: Bleeding, pain, infection, neurologic symptoms
Arm/Group | Serologic Arm
All-Cause Mortality (participants affected / at risk) | 0/292
Serious Adverse Events (participants affected / at risk) | 0/292
Other Adverse Events (participants affected / at risk) | 0/292

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT04383587/Prot_SAP_000.pdf